CLINICAL TRIAL: NCT03059810
Title: Clinical Evaluation of Investigational Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5903
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Participating Subjects (Experimental): Participating Subjects who are habitual soft contact lens wearers, aged 40 to 70 years of age, will be dispensed investigational contact lenses to be worn from 12-16 days, to include a total of 3 visits.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: etafilcon A — Investigational Contact Lens

SUMMARY:
3-visit dispensing study to evaluate the subjective feedback of a multifocal contact lens in a population of presbyopic patients. Subjects will wear the contact lenses for a total of 12-16 days.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Healthy adult males or females that are at least 40 years of age and no more than 70 years of age.
4. The subject must either be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not, respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".(Appendix B).
5. The subject is a current soft spherical or toric contact lens wearer (defined as a minimum of 6 hours of wear per day at least two days of the week for a minimum of 1 month prior to the study).
6. The subject's refractive spherical component must be between +1.25 Diopters (D) to +3.75 D in each eye.
7. The subject's refractive cylinder must be -1.00 D to -1.50 D in each eye.
8. The subject's refractive cylinder axis must be 90°±30° or 180°±30° in each eye.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
10. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.
11. The subject must have a wearable pair of spectacles if required for their distance vision.

Exclusion Criteria:

1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear.
2. Pregnancy or lactation.
3. Currently diagnosed with diabetes.
4. Infectious diseases (e.g. hepatitis, tuberculosis) or an immune-suppressive disease (e.g. HIV).
5. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
6. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
7. Any previous, or planned, ocular or intraocular surgery (e.g.radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), lid procedures, cataract surgery, retinal surgery, etc.).
8. A history of amblyopia, strabismus or binocular vision abnormality.
9. Any ocular infection or inflammation.
10. Any ocular abnormality that may interfere with contact lens wear.
11. Use of any ocular medication, with the exception of rewetting drops.
12. History of herpetic keratitis.
13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - EYE Center Optometric, Rocklin, California
  - Dr. Ted Brink & Associates, Jacksonville, Florida
  - Vistakon Research Clinic, Jacksonville, Florida
  - Golden Vision, Sarasota, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - University of Indiana School of Optometry, Bloomington, Indiana
  - Sacco Eye Group, Vestal, New York
  - Optometry Group, PLLC, Memphis, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 subjects were enrolled into this study. Of the enrolled subjects 63 were dispensed at least one study lens and 9 did not meet the eligibility criteria. All 63 dispensed subjects completed the study.
Groups:
- Etafilcon A With PVP: All subject wore the etafilcon A with PVP lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Etafilcon A With PVP
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etafilcon A With PVP
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 2
  White | 61
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 12-16 Day Follow-up
Population: Subjects that completed all visits without a major protocol deviation documented as impacted the assessment of the primary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Etafilcon A With PVP
Number analyzed (Participants) | 62
Units on a Scale | 47.33 (18.646)
Statistical Analysis 1: Comparison: Etafilcon A With PVP; It was a single arm study and the subjects' overall vision was compared against the baseline with the habitual lens. Sample size was determined using Power procedure in SAS 9.4 using the input from historical data (alpha=0.05); Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Linear mixed model (LMM); A 95% Confidence Interval for the least squares mean difference between the follow up and baseline was used to test for non-inferiority; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-4.6 to 5.9], Standard Deviation 2.63 — Mean difference was calculated as Test (at 12-16 days follow up) - Habitual (at baseline)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 2-weeks per subject.
Groups:
- Etafilcon A With PVP: All subjects wore the etafilcon A lens with PVP throughout the entire duration of the study.
Arm/Group | Etafilcon A With PVP
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03059810/Prot_SAP_000.pdf